CLINICAL TRIAL: NCT04506333
Title: Validation of the A&D UA-651 Oscillometric Blood Pressure Monitor in Children
Brief Title: Validation of A&D UA-651 in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Louisiana Monroe (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 1017
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2020-08-10 (Actual); Status verified 2020-08

CONDITIONS: Blood Pressure

STUDY DESIGN:
Intervention Model Description: The ISO/ESH/AAMI standards for validating blood pressure measurement devices will be used. In this model, participants' blood pressures are taken alternating between the test device and a reference device.
Masking Description: Investigators and assessors will need to know which device is associated with each measurement to perform analysis as specified in ISO/ESH/AAMI standards, but observers taking manual reference blood pressure measurements will be blinded as to each other's measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Small Cuff (Experimental): Participants with an upper-arm circumference of 6.3-9.4" may be placed in the small cuff arm.
  Interventions: Device: A&D UA-651 Blood Pressure Monitor; Device: ADC 740-N Manual Sphygmomanometer
- Medium Cuff (Experimental): Participants with an upper-arm circumference of 9.0-14.6" may be placed in the medium cuff arm.
  Interventions: Device: A&D UA-651 Blood Pressure Monitor; Device: ADC 740-N Manual Sphygmomanometer
- Lage Cuff (Experimental): Participants with an upper-arm circumference of 12.2-17.7" may be placed in the large cuff arm.
  The large cuff arm will use an adaptive study design. Per the AAMI/ESH/ISO standards, at least 1/6 of participants must fall into each cuff size arm for that cuff size, and of the participants assigned to each cuff size, at least 40% of those must fall in the upper and lower half of the cuff's size range. However, we do not anticipate many participants in our age range falling in the upper half of the large cuff size range (upper arm circumference > 14.95").
  Because of this, our plan is to validate the large cuff, but if enrolling a patient with a large cuff would require additional patients be enrolled to reach 1/6 of the total sample, the large cuff will be dropped from consideration and the validation completed with only the small and medium cuffs.
  Interventions: Device: A&D UA-651 Blood Pressure Monitor; Device: ADC 740-N Manual Sphygmomanometer

INTERVENTIONS:
Device: A&D UA-651 Blood Pressure Monitor — Test device to be validated.
Device: ADC 740-N Manual Sphygmomanometer — Reference device. Meets or exceeds ANSI/AAMI/ISO 81060-1 as required by ISO/ESH/AAMI standards.

SUMMARY:
This study will determine if the A&D UA-651 blood pressure monitor is valid in children.

ELIGIBILITY:
Inclusion Criteria:

* Parent permission
* Assent for participants aged 7-12
* Additional sequential selection criteria (described below)

Exclusion Criteria:

* Withdrawal of permission or assent
* Younger than 3 or older than 12 years of age
* Uncooperative participants, defined as refusing instructions from study personnel, coordinators, or observers
* Physical preclusion to taking blood pressure
* Participants who have any reference blood pressure measurement exceeding the 95th percentile plus 30mmHg for their age, sex, and height (urgent blood pressure level as defined by the American Academy of Pediatrics)
* Participants with systolic blood pressure difference of greater than 12mmHg or diastolic blood pressure difference of greater than 8mmHg between any two reference measurements

Sequential Selection Criteria:

Participants will be selected sequentially during study events. Per ISO/ESH/AAMI standards, participants must meet the following characteristics:

* at least 30% male and 30% female
* at least 1/6 using each of the three available cuff sizes (small, medium, large)
* for each cuff size, at least 40% in the upper half of the arm circumference range and at least 40% in the lower half of the arm circumference range.

If including a participant would require that additional participants be enrolled to meet the above criteria, that participant will not be included. For example, if only 2 small cuff participants are needed to complete the study, but a prospective participant would require a large cuff AND including that participant will require additional small or medium cuff participants to complete the study, then that prospective participant will not be included.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2020-08 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Blood Pressure Triplet | Immediate
  A valid set of 3 measurements (reference-test-reference) will be considered one outcome measurement for validation.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan J Donald, PharmD, Principal Investigator — University of Louisiana Monroe
Locations (1):
- University of Louisiana Monroe College of Pharmacy, Monroe, Louisiana, United States

REFERENCES:
- [Background] Stergiou GS, Palatini P, Asmar R, Ioannidis JP, Kollias A, Lacy P, McManus RJ, Myers MG, Parati G, Shennan A, Wang J, O'Brien E; European Society of Hypertension Working Group on Blood Pressure Monitoring. Recommendations and Practical Guidance for performing and reporting validation studies according to the Universal Standard for the validation of blood pressure measuring devices by the Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO). J Hypertens. 2019 Mar;37(3):459-466. doi: 10.1097/HJH.0000000000002039. PMID 30702492